CLINICAL TRIAL: NCT03262090
Title: Efficacy of Different Doses of Dexmedetomidine on the Prevention of Emergence Agitation in Children Undergoing Day Surgery With Desoflurane Anesthesia
Brief Title: Effect of Dexmedetomidine on the Prevention of Emergence Agitation in Children Undergoing Day Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Ying Jun She, MD, Dr., Guangzhou Women and Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YShe
Record Dates: First submitted 2017-08-18; First posted 2017-08-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Ambulatory Surgical Procedures
Keywords: Emergence Delirium; desoflurane; general anesthesia
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Aging

STUDY DESIGN:
Intervention Model Description: The aim of the present preliminary study was to determine the safety and efficacy of of intraoperative infusion of dexmedetomidine (DEX) that would prevent postoperative EA and ED in children undergoing day surgery with desoflurane anesthesia. Subjects who underwent day surgery were stratified into two age groups as follows: low to 3 years, and 3-9 years. Then they were randomly assigned to receive one of six doses of intravenous dexmedetomidine: 0,0.2, 0.4, 0.6, 0.8 ,1.0ug/kg before skin incision.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- control group (No Intervention): Subjects were randomly assigned to receive saline before skin incision
- 0.2ug/kg dexmedetomidine (Active Comparator): Subjects were randomly assigned to receive 0.2ug/kg intravenous dexmedetomidine before skin incision
  Interventions: Drug: 0.2ug/kg dexmedetomidine
- 0.4ug/kg dexmedetomidine (Active Comparator): Subjects were randomly assigned to receive 0.4ug/kg intravenous dexmedetomidine before skin incision
  Interventions: Drug: 0.4ug/kg dexmedetomidine
- 0.6ug/kg dexmedetomidine (Active Comparator): Subjects were randomly assigned to receive 0.6ug/kg intravenous dexmedetomidine before skin incision
  Interventions: Drug: 0.6ug/kg dexmedetomidine
- 0.8ug/kg dexmedetomidine (Active Comparator): Subjects were randomly assigned to receive 0.8ug/kg intravenous dexmedetomidine before skin incision
  Interventions: Drug: 0.8ug/kg dexmedetomidine
- 1.0ug/kg dexmedetomidine (Active Comparator): Subjects were randomly assigned to receive 1.0ug/kg intravenous dexmedetomidine before skin incision
  Interventions: Drug: 1.0ug/kg dexmedetomidine

INTERVENTIONS:
Drug: 0.2ug/kg dexmedetomidine — subjects were randomly assigned to receive 0.2ug/kg intravenous dexmedetomidine before skin incision
  Other Names: Age
  Arms: 0.2ug/kg dexmedetomidine
Drug: 0.4ug/kg dexmedetomidine — subjects were randomly assigned to receive 0.4ug/kg intravenous dexmedetomidine before skin incision
  Other Names: Age
  Arms: 0.4ug/kg dexmedetomidine
Drug: 0.6ug/kg dexmedetomidine — subjects were randomly assigned to receive 0.6ug/kg intravenous dexmedetomidine before skin incision
  Other Names: Age
  Arms: 0.6ug/kg dexmedetomidine
Drug: 0.8ug/kg dexmedetomidine — subjects were randomly assigned to receive 0.8ug/kg intravenous dexmedetomidine before skin incision
  Other Names: Age
  Arms: 0.8ug/kg dexmedetomidine
Drug: 1.0ug/kg dexmedetomidine — subjects were randomly assigned to receive 1.0ug/kg intravenous dexmedetomidine before skin incision
  Other Names: Age
  Arms: 1.0ug/kg dexmedetomidine

SUMMARY:
Emergence agitation/delirium (EA/ED) is a common complication in pediatric surgery patients, which increases the risk of developing postoperative airway obstruction and respiratory depression. In infants, there is a high incidence of emergence agitation (EA) after desoflurane anesthesia. The aim of the present preliminary study was to determine the safety and efficacy of of intraoperative infusion of dexmedetomidine (DEX) that would prevent postoperative EA and ED in children undergoing day surgery with desoflurane anesthesia

DETAILED DESCRIPTION:
subjects who underwent day surgery were stratified into two age groups as follows: low to 3 years group, and 3-12 years group. Then they were randomly assigned to receive one of six doses of intravenous dexmedetomidine: 0, 0.2, 0.4, 0.6, 0.8 ,1.0ug/kg before skin incision.

ELIGIBILITY:
Inclusion Criteria:

1. patients who undergo elective unilateral inguinal hernia or hydrocele testis day surgery
2. Patients who are American Society of Anesthesiologists classification I and II
3. Patients who are 4 months through 15 years of age

Exclusion Criteria:

1. children with history of respiratory tract infection 1 week preoperatively. 2. patients with preoperative liver and/or kidney dysfunction, or with mental abnormalities.

3. patients with any congenital malformation or acquired disease that could increase the risks of anesthesia and the dose of anesthetics (such as, but not limited to, congenital heart disease, hydronephrosis, nutrition dysplasia). 4. patients with long-term use of sedative or analgesic drugs.

Ages: 4 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 389 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
incidence of emergence agitation at different time interval after emergence | at 5min, 10min, 20min, 30min, 40min, 50min, 60min, 2h after emergence
  emergence agitation was evaluated by five-point scale

SECONDARY OUTCOMES:
sedation scales at different time interval after emergence | at 5min, 10min, 20min, 30min, 40min, 50min, 60min, 2h after emergence
  sedation was evaluated by MOAA/S scores
pain scale at different time interval after emergence | at 5min, 10min, 20min, 30min, 40min, 50min, 60min, 2h after emergence
  pain scale was evaluated by FLACC
incidence of emergence delirium at different time interval after emergence | at 5min, 10min, 20min, 30min, 40min, 50min, 60min, 2h after emergence
  emergence delirium was evaluated by five-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Xia Zheng, Doctor, Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children Medical Center, Guangzhou, Guangdong, China